CLINICAL TRIAL: NCT04899206
Title: ANGIOTENSIN AGENTS AND REDUCTION OF THE PRESCRIPTION OF ANTIDEPRESSANT DRUGS: A RETROSPECTIVE COHORT STUDY USING REAL-WORLD DATA
Status: Withdrawn | Type: Observational
Why Stopped: Lack of funding
Sponsor: Sebastian Videla (Other)
Collaborators: Institut d'Investigació Biomèdica de Bellvitge (Other); Institut Català de la Salut (Other)
Responsible Party: Sponsor-Investigator, Sebastian Videla, Head of the Clinical Research Support Unit, Hospital Universitari de Bellvitge
Organization: Hospital Universitari de Bellvitge (Other)
Other Study IDs: HUB-FC-2020-01
Record Dates: First submitted 2021-05-18; First posted 2021-05-24 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-06

CONDITIONS: ACE Inhibitors; ARB; Hypertension; Depression
Keywords: ACEI; ARB; ACE; RAS; Angiotension; Depression; Hypertension
MeSH Terms: conditions — Hypertension; Depression

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 38 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- ARBs only: Hypertensive patients under pharmacological treatment with ARBs
  Interventions: Drug: With an Antidepressant Drug; Drug: Without an Antidepressant Drug
- ACEIs only: Hypertensive patients under pharmacological treatment with ACEIs
  Interventions: Drug: With an Antidepressant Drug; Drug: Without an Antidepressant Drug
- ARBs + ACEIs: Hypertensive patients under pharmacological treatment with ARBs and ACEIs
  Interventions: Drug: With an Antidepressant Drug; Drug: Without an Antidepressant Drug
- Other Antihypertensive Drugs: Hypertensive patients under pharmacological treatment with non-angiotensin agents (diuretics, calcium channel blockers and/or β-blockers alone or combined among them)
  Interventions: Drug: With an Antidepressant Drug; Drug: Without an Antidepressant Drug
- Angiotensin Agents and Other Antihypertensive Drugs: Hypertensive patients under combined pharmacological treatment with Angiotensin Agents (ACEIs and/or ARBs) and Other Antihypertensives (non-angiotensin agents)
  Interventions: Drug: With an Antidepressant Drug; Drug: Without an Antidepressant Drug

INTERVENTIONS:
Drug: With an Antidepressant Drug — Current users of an antidepressant drug.
Drug: Without an Antidepressant Drug — Non-current users of an antidepressant drug.

SUMMARY:
A retrospective cohort study will be performed by analyzing data obtained from the Catalan Southern Metropolitan data warehouse system, which collects data from both hospitalized and primary care patients from the Bellvitge University Hospital's area of influence. The investigators will begin by gathering information only on patients treated with antihypertensive drugs, which then will be stratified in two groups: 1) Angiotensin Agents group; 2) Other Antihypertensive Agents (Non-Angiotensin Agents) group. Afterwards, a separated analysis will be performed to assess the effects of ARBs and ACEIs separately on the prescription of antidepressant drugs.

DETAILED DESCRIPTION:
Hypertension is a multifactorial disease and an important risk factor for cardiovascular and cerebrovascular diseases. Also, major depression is commonly found on these patients. Together, they represent a substantial burden for patients and their families, with an increased morbimortality and reduced life-quality. It also has a major social impact by increasing healthcare assistance demand and by affecting patients' daily-life productivity, therefore generating direct and indirect health-associated costs.

The Renin-Angiotensin System is one of the known pathways that modulate systemic and central nervous system inflammation. Basic research studies have shown ARBs-related allosteric changes on receptors implicated on the pathophysiology of schizophrenia and depression, and also a pharmacological reversal of depression-like behavior in rats after the administration of losartan. Human research studies have also presented evidence that points towards an antidepressant effect of some antihypertensive drugs.

A retrospective cohort study will be performed by analyzing data obtained from the Catalan Southern Metropolitan data warehouse system, which collects data from both hospitalized and primary care patients from the Bellvitge University Hospital's area of influence. The investigators will begin by gathering information only on patients treated with antihypertensive drugs, which then will be stratified in two groups: 1) Angiotensin Agents group; 2) Other Antihypertensive Agents (Non-Angiotensin Agents) group. Afterwards, a separated analysis will be performed to assess the effects of ARBs and ACEIs separately on the prescription of antidepressant drugs.

Our primary objective is to estimate the prevalence, incidence, and clearance (incidence of antidepressant drugs withdrawal) of antidepressant drugs prescription in hypertensive patients under treatment with angiotensin agents (ARBs and/or ACEIs).

Our secondary objectives are as follows:

I. For ARBs:

1. To estimate the prevalence of antidepressant drugs prescription in hypertensive patients under treatment with ARBs.
2. To estimate the clearance of antidepressant drugs prescription in patients concomitantly treated with ARBs and antidepressant drugs.
3. To estimate the incidence of antidepressant drugs initiation in patients with hypertension treated with ARBs.

II. For ACEIs:

1. To estimate the prevalence of antidepressant drugs prescription in hypertensive patients under treatment with ACEIs.
2. To estimate the clearance (incidence of antidepressant drugs withdrawal) of antidepressant drugs prescription in patients concomitantly treated with ACEIs and antidepressant drugs.
3. To estimate the incidence of antidepressant drugs initiation in patients with hypertension treated with ACEIs.

III. For other antihypertensive drugs (i.e., non-angiotensin agents: CCBs, β-blockers, and diuretics):

1. To estimate the prevalence of antidepressant drugs prescription in hypertensive patients under treatment with other antihypertensive drugs (non-angiotensin agents).
2. To estimate the clearance (incidence of antidepressant drugs withdrawal) of antidepressant drugs prescription in patients concomitantly treated with other antihypertensive drugs and antidepressant drugs.
3. To estimate the incidence of antidepressant drugs initiation in patients with hypertension treated with other antihypertensive drugs.

IV. To perform an exploratory comparative analysis among the different antihypertensive drugs sub-cohorts.

The protocol (Final Version: February 18th, 2021) was approved by the local Institutional Review Board (Ethic-and-Clinical-Investigation- Committee, code HUB-FC-2020-01, date April 20th, 2021). The study findings will be submitted to peer-reviewed journals and presented at relevant national and international scientific meetings.

ELIGIBILITY:
Inclusion Criteria:

* Patients that had an antihypertensive drug prescribed between January 1st, 2015 and December 31st, 2017, whose ATC codes can be obtained from the 'DATA WAREHOUSE' database
* Age ≥ 18 years old
* Both genders
* Patients with information available on the 'DATA WAREHOUSE' database
* Patients with a clinical visit or prescription done afterwards the date when the information for the study was last collected (this way we ensure that the patient included on the study remained alive after the end of the observation period)

Exclusion Criteria:

* Lack of information about the beginning of treatment with an antihypertensive and/or with an antidepressant drug.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients treated with antihypertensive drugs within the Bellvitge University Hospital's influence area (Barcelona's southern metropolitan area).
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2021-04-12 (Actual); Primary Completion 2021-12-20 (Actual); Study Completion 2025-12-20 (Estimated)

PRIMARY OUTCOMES:
Patients treated with antihypertensive drugs | 3 years
  Number of patients under treatment with antihypertensive drugs
Patients treated with an antidepressant drug | 3 years
  Number of patients under treatment with antidepressant drug

SECONDARY OUTCOMES:
Patients diagnosed with Hypertension | 3 years
  Number of patients diagnosed with Hypertension
Patients diagnosed with Depression | 3 years
  Number of patients diagnosed with Depression
Patients treated with ARBs | 3 years
  Number of patients treated with ARBs
Patients treated with ACEIs | 3 years
  Number of patients treated with ACEIs
Patients treated with other antihypertensive drugs | 3 years
  Number of patients treated with other antihypertensive drugs (i.e., non-ARBs and non-ACEIs).
Patients treated with Amitriptyline | 3 years
  Number of patients treated with Amitriptyline, since this is an antidepressant drug commonly used to treat neuropathic pain in our usual practice.
Patients treated with Duloxetine | 3 years
  Number of patients treated with Duloxetine, since this is an antidepressant drug commonly used to treat neuropathic pain in our usual practice.

CONTACTS AND LOCATIONS:
Overall Officials: Sebastián Videla, MD, PhD, Principal Investigator — Head of the Clinical Research Support Unit
Locations (1):
- Hospital Universitari de Bellvitge, L'Hospitalet de Llobregat, Catalonia, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Annerbrink K, Jonsson EG, Olsson M, Nilsson S, Sedvall GC, Anckarsater H, Eriksson E. Associations between the angiotensin-converting enzyme insertion/deletion polymorphism and monoamine metabolite concentrations in cerebrospinal fluid. Psychiatry Res. 2010 Sep 30;179(2):231-4. doi: 10.1016/j.psychres.2009.04.018. Epub 2010 May 16. PMID 20483169
- [Background] Aso E, Lomoio S, Lopez-Gonzalez I, Joda L, Carmona M, Fernandez-Yague N, Moreno J, Juves S, Pujol A, Pamplona R, Portero-Otin M, Martin V, Diaz M, Ferrer I. Amyloid generation and dysfunctional immunoproteasome activation with disease progression in animal model of familial Alzheimer's disease. Brain Pathol. 2012 Sep;22(5):636-53. doi: 10.1111/j.1750-3639.2011.00560.x. Epub 2012 Jan 13. PMID 22188425
- [Background] Bathina S, Das UN. Brain-derived neurotrophic factor and its clinical implications. Arch Med Sci. 2015 Dec 10;11(6):1164-78. doi: 10.5114/aoms.2015.56342. Epub 2015 Dec 11. PMID 26788077
- [Background] Borrajo A, Rodriguez-Perez AI, Diaz-Ruiz C, Guerra MJ, Labandeira-Garcia JL. Microglial TNF-alpha mediates enhancement of dopaminergic degeneration by brain angiotensin. Glia. 2014 Jan;62(1):145-57. doi: 10.1002/glia.22595. PMID 24272709
- [Background] Brownstein DJ, Salagre E, Kohler C, Stubbs B, Vian J, Pereira C, Chavarria V, Karmakar C, Turner A, Quevedo J, Carvalho AF, Berk M, Fernandes BS. Blockade of the angiotensin system improves mental health domain of quality of life: A meta-analysis of randomized clinical trials. Aust N Z J Psychiatry. 2018 Jan;52(1):24-38. doi: 10.1177/0004867417721654. Epub 2017 Jul 28. PMID 28754072
- [Background] Can A, Dao DT, Arad M, Terrillion CE, Piantadosi SC, Gould TD. The mouse forced swim test. J Vis Exp. 2012 Jan 29;(59):e3638. doi: 10.3791/3638. PMID 22314943
- [Background] Can A, Dao DT, Terrillion CE, Piantadosi SC, Bhat S, Gould TD. The tail suspension test. J Vis Exp. 2012 Jan 28;(59):e3769. doi: 10.3791/3769. PMID 22315011
- [Background] Cao YY, Xiang X, Song J, Tian YH, Wang MY, Wang XW, Li M, Huang Z, Wu Y, Wu T, Wu YQ, Hu YH. Distinct effects of antihypertensives on depression in the real-world setting: A retrospective cohort study. J Affect Disord. 2019 Dec 1;259:386-391. doi: 10.1016/j.jad.2019.08.075. Epub 2019 Aug 24. PMID 31470183
- [Background] Clark JD, Gebhart GF, Gonder JC, Keeling ME, Kohn DF. Special Report: The 1996 Guide for the Care and Use of Laboratory Animals. ILAR J. 1997;38(1):41-48. doi: 10.1093/ilar.38.1.41. No abstract available. PMID 11528046
- [Background] Deacon RM. Digging and marble burying in mice: simple methods for in vivo identification of biological impacts. Nat Protoc. 2006;1(1):122-4. doi: 10.1038/nprot.2006.20. PMID 17406223
- [Background] Farmer ME, Kittner SJ, Abbott RD, Wolz MM, Wolf PA, White LR. Longitudinally measured blood pressure, antihypertensive medication use, and cognitive performance: the Framingham Study. J Clin Epidemiol. 1990;43(5):475-80. doi: 10.1016/0895-4356(90)90136-d. PMID 2324788
- [Background] Goodman and Gilman's: The Pharmacological Basis of Therapeutics, 13th edition, New York: McGraw-Hill Medical, 2018.
- [Background] Grover MP, Ballouz S, Mohanasundaram KA, George RA, Sherman CD, Crowley TM, Wouters MA. Identification of novel therapeutics for complex diseases from genome-wide association data. BMC Med Genomics. 2014;7 Suppl 1(Suppl 1):S8. doi: 10.1186/1755-8794-7-S1-S8. Epub 2014 May 8. PMID 25077696
- [Background] Kessing LV, Rytgaard HC, Ekstrom CT, Torp-Pedersen C, Berk M, Gerds TA. Antihypertensive Drugs and Risk of Depression: A Nationwide Population-Based Study. Hypertension. 2020 Oct;76(4):1263-1279. doi: 10.1161/HYPERTENSIONAHA.120.15605. Epub 2020 Aug 24. PMID 32829669
- [Background] Kessing LV, Rytgaard HC, Gerds TA, Berk M, Ekstrom CT, Andersen PK. New drug candidates for depression - a nationwide population-based study. Acta Psychiatr Scand. 2019 Jan;139(1):68-77. doi: 10.1111/acps.12957. Epub 2018 Sep 4. PMID 30182363
- [Background] Komada M, Takao K, Miyakawa T. Elevated plus maze for mice. J Vis Exp. 2008 Dec 22;(22):1088. doi: 10.3791/1088. PMID 19229173
- [Background] Lenart L, Balogh DB, Lenart N, Barczi A, Hosszu A, Farkas T, Hodrea J, Szabo AJ, Szigeti K, Denes A, Fekete A. Novel therapeutic potential of angiotensin receptor 1 blockade in a rat model of diabetes-associated depression parallels altered BDNF signalling. Diabetologia. 2019 Aug;62(8):1501-1513. doi: 10.1007/s00125-019-4888-z. Epub 2019 May 3. PMID 31053872
- [Background] Li Z, Li Y, Chen L, Chen P, Hu Y. Prevalence of Depression in Patients With Hypertension: A Systematic Review and Meta-Analysis. Medicine (Baltimore). 2015 Aug;94(31):e1317. doi: 10.1097/MD.0000000000001317. PMID 26252317
- [Background] Lueptow LM. Novel Object Recognition Test for the Investigation of Learning and Memory in Mice. J Vis Exp. 2017 Aug 30;(126):55718. doi: 10.3791/55718. PMID 28892027
- [Background] Menendez E, Delgado E, Fernandez-Vega F, Prieto MA, Bordiu E, Calle A, Carmena R, Castano L, Catala M, Franch J, Gaztambide S, Girbes J, Goday A, Gomis R, Lopez-Alba A, Martinez-Larrad MT, Mora-Peces I, Ortega E, Rojo-Martinez G, Serrano-Rios M, Urrutia I, Valdes S, Vazquez JA, Vendrell J, Soriguer F. Prevalence, Diagnosis, Treatment, and Control of Hypertension in Spain. Results of the Di@bet.es Study. Rev Esp Cardiol (Engl Ed). 2016 Jun;69(6):572-8. doi: 10.1016/j.rec.2015.11.034. Epub 2016 Mar 12. English, Spanish. PMID 26979767
- [Background] Miller RE, Shapiro AP, King HE, Ginchereau EH, Hosutt JA. Effect of antihypertensive treatment on the behavioral consequences of elevated blood pressure. Hypertension. 1984 Mar-Apr;6(2 Pt 1):202-8. PMID 6724662
- [Background] Oliveira PA, Dalton JAR, Lopez-Cano M, Ricarte A, Morato X, Matheus FC, Cunha AS, Muller CE, Takahashi RN, Fernandez-Duenas V, Giraldo J, Prediger RD, Ciruela F. Angiotensin II type 1/adenosine A 2A receptor oligomers: a novel target for tardive dyskinesia. Sci Rep. 2017 May 12;7(1):1857. doi: 10.1038/s41598-017-02037-z. PMID 28500295
- [Background] Papp M, Willner P, Muscat R. An animal model of anhedonia: attenuation of sucrose consumption and place preference conditioning by chronic unpredictable mild stress. Psychopharmacology (Berl). 1991;104(2):255-9. doi: 10.1007/BF02244188. PMID 1876670
- [Background] Prut L, Belzung C. The open field as a paradigm to measure the effects of drugs on anxiety-like behaviors: a review. Eur J Pharmacol. 2003 Feb 28;463(1-3):3-33. doi: 10.1016/s0014-2999(03)01272-x. PMID 12600700
- [Background] Rygiel K. Can angiotensin-converting enzyme inhibitors impact cognitive decline in early stages of Alzheimer's disease? An overview of research evidence in the elderly patient population. J Postgrad Med. 2016 Oct-Dec;62(4):242-248. doi: 10.4103/0022-3859.188553. PMID 27763482
- [Background] Taura J, Valle-Leon M, Sahlholm K, Watanabe M, Van Craenenbroeck K, Fernandez-Duenas V, Ferre S, Ciruela F. Behavioral control by striatal adenosine A2A -dopamine D2 receptor heteromers. Genes Brain Behav. 2018 Apr;17(4):e12432. doi: 10.1111/gbb.12432. Epub 2017 Nov 17. PMID 29053217
- [Background] Williams LJ, Pasco JA, Kessing LV, Quirk SE, Fernandes BS, Berk M. Angiotensin Converting Enzyme Inhibitors and Risk of Mood Disorders. Psychother Psychosom. 2016;85(4):250-2. doi: 10.1159/000444646. Epub 2016 May 27. No abstract available. PMID 27230871